CLINICAL TRIAL: NCT03592329
Title: Brain Mechanisms of Vagus Nerve Stimulation and Stress Reduction Training for Migraine
Brief Title: Vagus Nerve Stimulation and Stress Reduction Training for Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Vitaly Napadow, Ph.D., Lic.Ac., Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2018P001184; P01AT009965 (NIH)
Record Dates: First submitted 2018-05-24; First posted 2018-07-19 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- active tVNS + SRT A (Experimental): active tVNS and Stress Reduction Training A
  Interventions: Behavioral: Stress Reduction Training A; Device: active tVNS
- active tVNS + SRT B (Experimental): active tVNS and Stress Reduction Training B
  Interventions: Device: active tVNS; Behavioral: Stress Reduction Training B
- sham tVNS + SRT A (Other): sham stimulation and Stress Reduction Training A
  Interventions: Behavioral: Stress Reduction Training A; Device: sham tVNS
- sham tVNS + SRT B (Other): sham tVNS and Stress Reduction Training B
  Interventions: Behavioral: Stress Reduction Training B; Device: sham tVNS

INTERVENTIONS:
Behavioral: Stress Reduction Training A — twice weekly "booster" sessions and weekly instructor-led sessions for 8 weeks plus home practice sessions
  Other Names: SRT A
  Arms: active tVNS + SRT A; sham tVNS + SRT A
Device: active tVNS — non-painful electrical stimulation of the auricle
  Other Names: transcutaneous vagus nerve stimulation
  Arms: active tVNS + SRT A; active tVNS + SRT B
Behavioral: Stress Reduction Training B — twice weekly "booster" sessions and weekly instructor-led sessions for 8 weeks plus home practice sessions
  Other Names: SRT B
  Arms: active tVNS + SRT B; sham tVNS + SRT B
Device: sham tVNS — sham stimulation
  Arms: sham tVNS + SRT A; sham tVNS + SRT B

SUMMARY:
This study design has two components: 1) a cross-sectional assessment of brain activity and inflammation in migraine patients compared to healthy controls and 2) an assessment of 8 weeks of a combination therapy approach to treating migraine.

DETAILED DESCRIPTION:
Chronic pain is the most prevalent and disabling medical condition, and no single therapy has proven to be completely successful for alleviating pain, such as migraine headache. It is well documented, and recommended in the recent Institute of Medicine (IOM) report, that a multimodal approach is optimal for pain management. This study will evaluate a combination transcutaneous vagus nerve stimulation and stress reduction training for migraine.

Investigators will recruit participants who have migraines and randomize to one of four potential treatment arms (real or sham stimulation + real or sham stress reduction training). Brain imaging (MRI and PET) and clinical data will be collected before and after 8 weeks of the combination therapy.

Healthy controls will also be recruited for collection of the same baseline brain imaging and clinical data, but with no treatment or second data collection phase.

Findings from this research will help elucidate brain activity and inflammation associated with migraines and evaluate the efficacy of the combination therapy in reducing migraine.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be between 18 and 65 years of age.
2. Migraine Diagnosis and general health otherwise.
3. Willingness to attend twice- weekly treatment session at Cambridge Health Alliance for 8 weeks.
4. Able to give written consent and participate in group interventions in English.

Healthy Volunteers between the ages of 18 and 65 can participate in this study.

Exclusion Criteria:

1. Major illness, psychiatric condition, or neurological disease.
2. Previous experience with stress reduction training (such as mindfulness training, MBSR, MBCT, Relaxation Response) or more than 15 home mediation practice sessions in the past month, or more than 10 classes in yoga, Tai Chi, or Qi Gong in the past 3 months
3. Any condition that would prohibit MRI scanning

Healthy Volunteers have the same eligibility constraints with the addition of current or past history of migraine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Brain activity changes in migraine patients in response to treatment | 8 weeks post treatment
  fMRI BOLD signal (percent BOLD signal change) from baseline to post-treatment, compared across treatment groups.
Brain inflammation changes in migraine patients in response to treatment | 8 weeks post treatment
  PET [11C]PBR28 signal, quantified as Standardized Uptake Value Ratio (SUVR; i.e., tissue radioactivity / injected dose / weight) change from baseline to post-treatment, compared across treatment groups for migraine patients.

SECONDARY OUTCOMES:
Brain activity differences between Migraine patients and healthy controls | 3 weeks
  fMRI BOLD signal differences (percent BOLD signal change) between group maps for migraine patients and healthy controls at baseline
Brain inflammation differences between Migraine patients and healthy controls | 3 weeks
  PET [11C]PBR28 signal, quantified as Standardized Uptake Value Ratio (SUVR; i.e., tissue radioactivity / injected dose / weight), differences between healthy controls and migraine patients at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Napadow, PhD,Lic.Ac., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Anthinoula A. Martinos Center, Charlestown, Massachusetts, United States

DOCUMENTS (1):
  • Informed Consent Form (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT03592329/ICF_000.pdf